CLINICAL TRIAL: NCT06926595
Title: Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) With Low-Dose Post-Transplant Cyclophosphamide for Prophylaxis of Graft-versus-Host Disease in Hematological Malignancies
Brief Title: Allogeneic HSCT With Low-Dose Post-Transplant Cyclophosphamide for GVHD Prevention
Acronym: GVHD-PTCy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Cioccio, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-24-047; PSCI-24-047 (Other: Penn State Cancer Institute)
Record Dates: First submitted 2025-04-10; First posted 2025-04-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Graft-versus-Host Disease (GVHD); Hematologic Malignancies; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, Phase 2 clinical trial. All participants will receive the same intervention, which is low-dose (25 mg/kg) post-transplant cyclophosphamide (PTCy) for GVHD prophylaxis, in combination with tacrolimus and mycophenolate mofetil (MMF). The study will assess the safety and efficacy of this regimen in patients undergoing allogeneic stem cell transplantation using peripheral blood stem cells from matched sibling, matched unrelated, and haploidentical donors, following reduced-intensity or non-myeloablative conditioning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-Dose PTCy for GVHD Prophylaxis (Experimental): Participants in this single-arm study will receive low-dose (25 mg/kg) post-transplant cyclophosphamide (PTCy) on days +3 and +4 following allogeneic hematopoietic stem cell transplantation. This will be administered in combination with tacrolimus and mycophenolate mofetil (MMF) for graft-versus-host disease (GVHD) prophylaxis. The study includes patients receiving transplants from matched sibling, matched unrelated, single allelic mismatched unrelated, and haploidentical donors following reduced-intensity or non-myeloablative conditioning.
  Interventions: Drug: Cyclophosphamide (primary intervention for GVHD prophylaxis)

INTERVENTIONS:
Drug: Cyclophosphamide (primary intervention for GVHD prophylaxis) — This study evaluates the use of low-dose (25 mg/kg) post-transplant cyclophosphamide (PTCy) for prophylaxis of Graft-versus-Host Disease (GVHD) following allogeneic stem cell transplantation. The intervention involves administering PTCy on days +3 and +4 post-transplant, in combination with tacrolimus and mycophenolate mofetil (MMF) for GVHD prevention. The goal is to assess the safety and efficacy of this regimen in patients undergoing reduced-intensity or non-myeloablative conditioning using peripheral blood stem cells from matched sibling, matched unrelated, and haploidentical donors
  Other Names: Tacrolimus (part of the GVHD prophylaxis regimen); Mycophenolate mofetil (MMF) (part of the GVHD prophylaxis regimen)

SUMMARY:
This Phase 2, single-arm, open-label study aims to evaluate the safety and efficacy of low-dose (25 mg/kg) post-transplant cyclophosphamide (PTCy) for prophylaxis of Graft-versus-Host Disease (GVHD) in patients undergoing allogeneic stem cell transplantation following reduced-intensity or non-myeloablative conditioning. The study will focus on matched sibling, matched unrelated, and haploidentical peripheral blood stem cell donors. The primary endpoint is 1-year GVHD-Free Relapse-Free Survival (GRFS). The study seeks to determine if low-dose PTCy offers similar outcomes as higher doses, with potentially reduced toxicity.

DETAILED DESCRIPTION:
This study investigates the use of low-dose post-transplant cyclophosphamide (PTCy) for GVHD prophylaxis in a Phase 2, single-arm design. It involves patients receiving allogeneic stem cell transplantation with peripheral blood stem cells from matched sibling, matched unrelated, and haploidentical donors, following reduced-intensity or non-myeloablative conditioning. The aim is to evaluate 1-year GVHD-Free Relapse-Free Survival (GRFS) using 25 mg/kg of PTCy administered on days +3 and +4, in combination with tacrolimus and mycophenolate mofetil (MMF).

The study builds on previous research that has shown the effectiveness of PTCy in preventing GVHD in various transplant settings, including haploidentical and matched unrelated donors. Lower doses of PTCy, such as 25 mg/kg, have been shown to be effective in other settings with reduced toxicity compared to the standard 50 mg/kg dose, and this study will assess whether the same holds true for peripheral blood stem cell transplants.

The findings from this trial will help determine the optimal dosing strategy for PTCy in GVHD prophylaxis, with the potential to improve patient outcomes by minimizing toxicity while maintaining efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older at the time of study enrollment.
* Patients with acute leukemia (acute myeloid leukemia, acute lymphoblastic leukemia, mixed phenotype acute leukemia) or chronic myeloid leukemia with no circulating blasts and less than 5% blasts in the bone marrow.

Flow cytometric, polymerase chain reaction (PCR) or next generation sequencing (NGS) detected measurable residual disease is permitted.

* Patients with myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia with no circulating blasts and less than 10% blasts in the bone marrow (exception allowed due to lack of difference in outcomes with <5% vs 5-10% blasts in this disease).
* Patients with secondary acute myeloid leukemia progressing from pre-existing myelodysplastic syndrome, myeloproliferative disease (MPN), or MDS/MPN overlap syndrome.
* Patients with relapsed or refractory chronic lymphocytic leukemia/small lymphocytic lymphoma who are indicated for allogeneic stem cell transplantation.
* Patients with lymphoma who are indicated for allogeneic stem cell transplantation, including follicular lymphoma, Hodgkin lymphoma, diffuse large B cell lymphoma (including primary mediastinal B cell lymphoma), mantle cell lymphoma, peripheral T cell lymphomas, and Richter's transformation.
* Planned reduced intensity or non-myeloablative conditioning regimen.
* Patients must have a related or unrelated peripheral blood stem cell donor as follows:

Sibling donor must be at least haploidentical using high resolution DNA-based HLA typing.

Children or parent donor must be at least haploidentical using high resolution DNA-based HLA typing. Children donors must be at least 18 years of age at the time of evaluation.

Unrelated donors must be a 7/8 or 8/8 match at HLA-A, B, C, and DRB1 at high resolution using DNA based typing.

* Cardiac function: must demonstrate at ejection fraction of at least 40%.
* Pulmonary function: must have FEV1 of at least 50% predicted, and DLCO corrected for hemoglobin of at least 40% predicted.
* Karnofsky performance status at least 70%.
* Women of childbearing potential (WOCP), defined as not surgically sterile (hysterectomy, tubal ligation, or oophorectomy) or at least 1 year postmenopausal, must have a negative serum pregnancy test before conditioning regimen.
* Female patients (unless post-menopausal or surgically sterilized) must agree to practice two effective methods of contraception simultaneously or agree to completely abstain from heterosexual intercourse from the time of signing informed consent through 12 months post-transplant.
* Male patients (even if surgically sterilized) who are partners of women of childbearing potential must agree to practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant.

Exclusion Criteria:

* Prior allogeneic stem cell transplant.
* Active central nervous system (CNS) involvement by malignant cells.
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication with progression or no clinical improvement).
* Seropositive for human immunodeficiency virus (HIV) with detectable viral load, hepatitis B virus (HBV) or hepatitis C virus (HCV) with detectable viral load. Hepatitis B surface antibody positive due to vaccination or natural immunity are permitted. Patients previously treated for HCV and considered to be in sustained virologic remission (SVR) are allowed.
* Myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III-IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
* Pregnant or lactating female patients (unless feeding via formula). Women of childbearing potential (WOCBP) are required to have a negative serum or urine pregnancy test prior to conditioning regimen.
* Serious medical or psychiatric illness likely to interfere with participation in the study.
* Use of investigational agents.
* Haploidentical related recipient who are positive for DSA ≥ 5000 MFI by solid phase microarray method (Luminex).
* Any patient with steroid dose more than 10 mg/day within a week of registration.
* Autoimmune disorder requiring any active immunosuppression therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Without Grade III/IV Acute Graft-Versus-Host Disease (GVHD) at 1 Year | 1 year post-transplant
  The number of subjects without Grade III/IV acute graft-versus-host disease (GVHD) at one year following allogeneic stem cell transplantation, assessed using the Modified Glucksberg Criteria (Grade III: severe organ involvement, e.g., skin stage 3-4, liver or gut stage 2-3; Grade IV: life-threatening dysfunction, e.g., skin, liver, or gut stage 4).
Number of Subjects Without Chronic Graft-Versus-Host Disease (GVHD) Requiring Systemic Treatment at 1 Year | 1 year post-transplant
  The number of subjects without chronic graft-versus-host disease (GVHD) requiring systemic treatment (e.g., corticosteroids or immunosuppressive therapy) at one year following allogeneic stem cell transplantation with low-dose post-transplant cyclophosphamide (25 mg/kg), assessed per the NIH Consensus Criteria for chronic GVHD.
Number of Subjects Without Relapse or Disease Progression at 1 Year | 1 year post-transplant
  The number of subjects without relapse or disease progression at one year following allogeneic stem cell transplantation, defined as the reappearance of the underlying disease or worsening of disease burden, assessed by standard clinical and laboratory measures (e.g., bone marrow biopsy, or disease-specific markers such as minimal residual disease [MRD] testing) per the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cioccio, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be published in a peer-reviewed journal.